CLINICAL TRIAL: NCT03915964
Title: A Randomized, Active-Controlled, Parallel-Group, Phase 3b/4 Study of Baricitinib in Patients With Rheumatoid Arthritis
Brief Title: A Study of Baricitinib (LY3009104) in Participants With Rheumatoid Arthritis
Acronym: RA-BRIDGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17172; I4V-MC-JAJA (Other: Eli Lilly and Company); 2018-003351-37 (EudraCT Number)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib; Tumor Necrosis Factor Inhibitors; Etanercept; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Baricitinib Low Dose (Experimental): Baricitinib administered orally.
  Interventions: Drug: Baricitinib
- Baricitinib High Dose (Experimental): Baricitinib administered orally.
  Interventions: Drug: Baricitinib
- TNF Inhibitor (Active Comparator): Adalimumab or etanercept administered subcutaneously (SC) per standard of care.
  Interventions: Drug: TNF Inhibitor

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
  Arms: Baricitinib High Dose; Baricitinib Low Dose
Drug: TNF Inhibitor — Administered SC
  Other Names: Etanercept; Adalimumab
  Arms: TNF Inhibitor

SUMMARY:
This post-marketing study is designed to compare the safety of baricitinib versus tumor necrosis factor (TNF) inhibitors with respect to venous thromboembolic events (VTEs) when given to participants with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have at least one of the following characteristics:

  * Documented evidence of a VTE prior to this study
  * At least 60 years of age
  * A body mass index (BMI) greater than or equal to 30 kilograms per meter squared (kg/m²), or
  * Age 50 to less than 60 years and BMI 25 to less than 30 kg/m².
* Participants must have an inadequate response or intolerance to at least 1 disease-modifying antirheumatic drugs (DMARD) (synthetic or biologic).

Exclusion Criteria:

* Participant should have no reason to not take a TNF inhibitor.
* Participants must not be pregnant or breastfeeding.
* Participants must not have had more than one VTE.
* Participants must not have cancer.
* Participants must not have active herpes zoster, serious infection, active tuberculosis, or any other serious illness.
* Participants must not have had a live vaccine within four weeks of study start.
* Participants must not have participated in any other clinical trial within four weeks of study start.
* Participants must not have a history of IV drug use, other illicit drug abuse, or chronic alcohol abuse in the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2663 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Time from First Dose of Study Treatment to First Event of Venous Thromboembolism (VTE) | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First Event of VTE

SECONDARY OUTCOMES:
Time from First Dose of Study Treatment to First Arterial Thromboembolic Event (ATE) | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First ATE
Time from First Dose of Study Treatment to First Major Adverse Cerebro-Cardiovascular Event (MACE) | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First MACE
Time from First Dose of Study Treatment to First Malignancy (excluding nonmelanoma skin cancer [NMSC]) | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First Malignancy (excluding NMSC)
Time from First Dose of Study Treatment to First Opportunistic Infection | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First Opportunistic Infection
Time from First Dose of Study Treatment to First Serious Infection | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First Serious Infection

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (261):
- United States (81):
  - Arizona Arthritis & Rheumatology Research, PLLC, Flagstaff, Arizona
  - Arthrocare, Arthritiscare & Research Pc, Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - Hope Research Institute, Peoria, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Tucson, Arizona
  - Medvin Clinical Research - Covina, Covina, California
  - St Joseph Heritage Healthcare, Fullerton, California
  - Christine Thai, MD, Huntington Beach, California
  - Private Practice - Dr. Christine J. Leehealey, Irvine, California
  - Desert Medical Advances, Rancho Mirage, California
  - Rheumatology Center of San Diego, San Diego, California
  - East Bay Rheumatology Medical Group, Inc, San Leandro, California
  - Dan La, MD Inc, Tujunga, California
  - Robin K. Dore MD, Inc, Tustin, California
  - Inland Rheumatology & Osteoporosis Medical Group, Upland, California
  - Medvin Clinical Research - Weidmann, Van Nuys, California
  - Medvin Clinical Research - Whittier, Whittier, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Rheumatology Associates of South Florida, Boca Raton, Florida
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - IRIS Research and Development, LLC, Plantation, Florida
  - Qps-Mra, Llc, South Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Arthritis & Rheumatology of Georgia, Atlanta, Georgia
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - St. Luke's Intermountain Research Center, Boise, Idaho
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Qualmedica Research, LLC, Evansville, Indiana
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Center for Arthritis and Osteoporosis, Elizabethtown, Kentucky
  - Accurate Clinical Research, Lake Charles, Louisiana
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - University of Michigan, Brighton, Michigan
  - West Michigan Rheumatology, Grand Rapids, Michigan
  - Advanced Rheumatology, PC, Okemos, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Westroads Clinical Research, Inc., Omaha, Nebraska
  - Allied Clinical Research, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Santa Fe Rheumatology, Santa Fe, New Mexico
  - Accellacare - Charlotte, Charlotte, North Carolina
  - M3-Emerging Medical Research, LLC, Durham, North Carolina
  - Piedmont Rheumatology, P.A., Hickory, North Carolina
  - Cape Fear Arthritis Care, Leland, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Cincinnati Rheumatic Disease Study Group, Cincinnati, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, Bethlehem, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading,LLC, Wyomissing, Pennsylvania
  - Pennsylvania Regional Center for Arthritis and Osteoporosis Research, Wyomissing, Pennsylvania
  - Regional Health Clinical Research, Rapid City, South Dakota
  - Accurate Clinical Management, Baytown, Texas
  - Arthritis & Osteoporosis Clinic of Brazos Valley, College Station, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Accurate Clinical Management - Houston, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Research Physicians Network, LLC, Houston, Texas
  - Accurate Clinical Research, League City, Texas
  - Accurate Clinical Research, Inc., San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Accurate Clinical Management, Sugar Land, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Tomball, Texas
  - DM Clinical Research/Rheumatology Clinic of Houston, Tomball, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
  - The Vancouver Clinic, Vancouver, Washington
  - CAMC Health Education and Research Institute Inc, Charleston, West Virginia
- Australia (5):
  - Optimus Clinical Research, Botany, New South Wales
  - Genesis Research Services, Newcastle, New South Wales
  - Rheumatology Research Unit, Maroochydore, Queensland
  - Southern Clinical Research, Hobart, Tasmania
  - Emeritus Research, Camberwell, Victoria
- Austria (3):
  - Medizinische Universität Wien, Vienna, Vienna
  - Wilhelminenspital, Vienna, Vienna
  - Rheuma-Zentrum Oberlaa GmbH, Vienna
- Belgium (3):
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels, Bruxelles-Capitale, Région de
  - ZNA Jan Palfijn, Merksem, Flanders
  - Reuma Clinic, Locatie Jaarbeurslaan, Genk, Limburg
- Czechia (13):
  - Revmacentrum MUDr. Mostera, s.r.o., Brno, Brno-město
  - Revmatologie.s.r.o., Brno, Brno-město
  - Artroscan, s.r.o., Ostrava, Moravskoslezský kraj
  - INREA s.r.o., Ostrava, Ostrava Město
  - ARTHROHELP s.r.o., Pardubice, Pardubický kraj
  - Clintrial s.r.o., Prague, Praha 10
  - Revmatologie MUDr. Štejfová, Prague, Praha 4
  - Revmatologicky ustav, Prague, Praha, Hlavní Mešto
  - REVMACLINIC s.r.o., Brno, South Moravian
  - Medical Plus, Uherské Hradiště, Zlín
  - PV Medical Services s.r.o., Zlín, Zlín
  - Revmatologicka ambulance, Prague
  - Affidea Praha, s.r.o., Prague
- Denmark (2):
  - Regionshospitalet Silkeborg, Silkeborg, Central Jutland
  - Reumatologisk Ambulatorie, Svendborg Hospital Odense Universitet Hospital, Svendborg, Region Syddanmark
- France (12):
  - CHU de Nice, Nice, Alpes-Maritimes
  - CHU Strasbourg-Hautepierre, Strasbourg, Alsace
  - Bordeaux University Hospital - Pellegrin, Bordeaux, Aquitaine
  - Hôpital Edouard Herriot, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Regional D'Orleans, Orléans, Centre-Val de Loire
  - Hôpital Pierre-Paul Riquet, Toulouse, Haute-Garonne
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes, Loire-Atlantique
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHD Vendee, La Roche-sur-Yon, Vendée
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Roger Salengro, Lille
  - Pitie Salpetriere University Hospital, Paris
- Germany (9):
  - CIRI- Center of Innovative Diagnostics and Therapeutics Rheumatology/Immunology, Frankfurt am Main, Hesse
  - Rheumazentrum Prof.Neeck MVZ, Bad Doberan, Mecklenburg-Vorpommern
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Rheumazentrum Ratingen Studienambulanz, Ratingen, North Rhine-Westphalia
  - Institut für Präventive Medizin & Klinische Forschung GbR, Magdeburg, Saxony-Anhalt
  - Praxis für Rheumatologie und Innere, Berlin
  - Schlosspark Klinik, Berlin
  - HRF II - Hamburger Rheuma Forschungszentrum II MVZ für Rheumatologie und Autoimmunmedizin Hamburg GmbH / -T, Hamburg
  - Hamburger Rheuma Forschungszentrum I / Dres Raabe & Heintz, Hamburg
- Greece (3):
  - Attikon General University Hospital, Chaïdári, Attikí
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki, Kentrikí Makedonía
  - University Hospital of Alexandroupolis, Alexanroupolis, Évros
- Hungary (6):
  - CRU Hungary Kft., Miskolc, Borsod-Abauj Zemplen county
  - Revita Clinic, Budapest, Pest County
  - Clinexpert Kft., Budapest, Pest County
  - Vital Medical Center, Veszprém, Veszprém City
  - Debreceni Egyetem - Kenézy Gyula Egyetemi Oktatókórház, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- Israel (7):
  - Meir Medical Center, Kfar Saba, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Barzilai Medical Center, Ashkelon, Southern District
  - Sourasky Medical Center, Tel Aviv, Tell Abīb
  - Rambam Health Care Campus, Haifa, Ḥeifā
  - Carmel Hospital, Haifa, Ḥeifā
  - Bnai Zion Medical Center, Haifa, Ḥeifā
- Italy (6):
  - Clinical Research Center - Universita Degli Studi Gabriele d'Annunzio, Chieti, Abruzzo
  - Ospedale Luigi Sacco, Milan, Milano
  - Ospedale Le Scotte, Siena, Tuscany
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - University of Campania Luigi Vanvitelli, Napoli
  - Policlinico GB Rossi Borgo Roma, Verona
- Lithuania (3):
  - Republican Hospital of Kaunas, Kaunas, Kauno Miestas
  - Centro poliklinika, Vilnius
  - Respublikin Šiauli ligonin, Šiauliai, Šiauliai County
- Netherlands (2):
  - PT&R / PreCare Trial & Recruitment, Born, Limburg
  - Medische Centrum Leeuwarden, Leeuwarden, Provincie Friesland
- Poland (18):
  - Ai Centrum Medyczne Sp. Z O.O., Poznan, Greater Poland Voivodeship
  - Prywatna Praktyka Lekarska Prof. UM dr hab. med. Pawel Hrycaj, Poznan, Greater Poland Voivodeship
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Klinika Reumatologii i Ukladowych Chorób Tkanki Lacznej, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun, Torun, Kuyavian-Pomeranian Voivodeship
  - Samodzielny Publiczny Zespol Opieki Zdrowotnej W Tomaszowie Lubelskim, Tomaszów Lubelski, Lublin Voivodeship
  - Twoja Przychodnia Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - NZOZ Lecznica MAK-MED s.c., Nadarzyn, Masovian Voivodeship
  - Medycyna Kliniczna, Warsaw, Masovian Voivodeship
  - Rheuma Medicus- Zak��ad Opieki Zdrowotnej, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park, Warsaw, Masovian Voivodeship
  - ETG Warszawa, Warsaw, Masovian Voivodeship
  - Centrum Medyczne AMED Warszawa Targowek, Warsaw, Masovian Voivodeship
  - Osteo Medic sc A. Racewicz, J. Supronik, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - BIF-MED, Bytom, Silesian Voivodeship
  - Centrum Medyczne Pratia Katowice, Katowice, Silesian Voivodeship
  - Slaskie Centrum Reumatologii, Rehabilitacji I Zapobiegania Niepelnosprawnosci Im. Gen.J.Zietka, Ustroń, Silesian Voivodeship
  - Ambulatorium Barbara Bazela, Elblag, Warmian-Masurian Voivodeship
- Puerto Rico (5):
  - Centro Reumatologico Caguas, Caguas
  - Ponce Medical School Foundation Inc., Ponce
  - Latin Clinical Trial Center, San Juan
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
  - Mindful Medical Research, San Juan
- Romania (9):
  - C.M.D.T.A. Neomed, Brasov, Brașov County
  - Cmi Cristei Dorica, Brăila, Brăila County
  - Spital Clinic Sf. Maria, Bucharest, București
  - Delta Health Care, Bucharest, București
  - CCBR Clinical Research, Bucharest, București
  - Spitalul Clinic Judetean de Urgenta Sf. Apostol Andrei, Galati, Galați County
  - RK Medcenter, Iași, Iaşi
  - Spitalul Judeean de Urgen Dr. Constantin Opri Baia Mare, Baia Mare, Maramureş
  - Sc Medaudio-Optica Srl, Râmnicu Vâlcea, Vâlcea County
- Russia (15):
  - Kursk Regional Clinical Hospital, Kursk, Kursk Oblast
  - Gbuz Lokb, Saint-Petersburg, Leningradskaya Oblast'
  - Moscow Clinical Research Center, Moscow, Moscow
  - Federal State Budgetary Scientific Institution Research Institute Rheumatology named after V.A.Nasonova, Moscow, Moscow
  - M. F. Vladimirskiy Moscow Regional Research Clinical Institute, Moscow, Moscow
  - First Moscow State Medical University I.M. Sechenov, Moscow, Moscow Oblast
  - Nizhny Novgorod City Clinical Hospital Number 5, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Ryazan Regional Clinical Cardiological Dispensary, Ryazan, Ryazan Oblast
  - Clinical Rheumatology hospital #25, Saint Petersburg, Sankt-Peterburg
  - North-Western State Medical University named after I.I.Mechnikov, Saint Petersburg, Sankt-Peterburg
  - Tula Regional Clinical Hospital, Tula, Tula Oblast
  - GUZ UOKB, Ulyanovsk, Ulyanovsk Oblast
  - Karelia Republican Hospital V.A. Baranova, Petrozavodsk
  - Regional Clinical Hospital of the Saratov Region, Saratov
  - Research & Practice, Yaroslavl
- Slovakia (6):
  - ALBAMED s.r.o., Zvolen, Banská Bystrica Region
  - ROMJAN s.r.o., Bratislava, Bratislava Region
  - Artromac n.o., Košice, Košice Region
  - REUMED s.r.o., Spišská Nová Ves, Košice Region
  - LERAM s.r.o., Topoľčany, Nitra Region
  - Reumacentrum s.r.o., Partizánske, Trenčín Region
- South Africa (9):
  - Netcare Greenacres Hospital, Port Elizabeth, Eastern Cape
  - FARMOVS, Bloemfontein, Free State
  - Iatros International, Bloemfontein, Free State
  - Clinresco Centres, Kempton Park, Gauteng
  - University of Pretoria - Faculty of Health Sciences, Pretoria, Gauteng
  - Precise Clinical Solutions, Chatsworth, KwaZulu-Natal
  - Netcare Umhlanga Hospital, Umhlanga, KwaZulu-Natal
  - Arthritis Clinical Trial Centre, Cape Town, Western Cape
  - Winelands Medical Research Centre, Stellenbosch, Western Cape
- Spain (21):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [La Coruña]
  - Clínica Gaias - Santiago, Santiago de Compostela, A Coruña [La Coruña]
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Osi Bilbao-Basurto, Bilbao, Basque Country
  - Clínica Sagrada Familia, Barcelona, Catalunya [Cataluña]
  - Hospital Quiron Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Corporació Sanitària Parc Taulí, Sabadell, Catalunya [Cataluña]
  - Consorci Sanitari Integral. Hospital Moisés Broggi, Sant Joan Despí, Sant Joan Despí, Catalunya [Cataluña]
  - Hu Reina Sofia, Córdoba, Córdoba
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, Galicia [Galicia]
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid, Comunidad de
  - Hospital Universitario Getafe, Getafe, Madrid, Comunidad de
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Comunidad de
  - CHUVI- Hospital do Meixoeiro, Vigo, Pontevedra [Pontevedra]
  - Hospital Quirónsalud Córdoba, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Quiron Infanta Luisa, Seville
- Switzerland (3):
  - University Hospital Basel, Basel, Canton of Basel-City
  - Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - HFR Fribourg - Hôpital Cantonal, Fribourg
- Turkey (Türkiye) (6):
  - Eskisehir Osmangazi University, Eskişehir, Eskişehir
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi, Stanbul, Istanbul
  - Trakya University, Edirne
  - Istanbul University Cerrahpasa Medical School Internal Diseases Institute, Istanbul
  - Izmir Katip Celebi Ataturk Egitim Arastirma Hastanesi, Izmir
  - Necmettin Erbakan Meram Medical Fac., Konya
- United Kingdom (14):
  - Christchurch Hospital, Christchurch, Bournemouth
  - Derriford Hospital, Plymouth, Devon
  - Torbay Hospital, Torquay, Devon
  - The Dudley Group NHS Foundation Trust, Dudley, England
  - Royal Free London NHS Foundation Trust, London, England
  - The Royal Cornwall Hospital, Truro, England
  - Mid Essex Hospital Services NHS Trust, Chelmsford, Essex
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - Hull and East Yorkshire Hospitals NHS Trust, Hull, Kingston Upon Hull
  - Northumbria Healthcare NHS Foundation Trust, Newcastle upon Tyne, North Tyneside
  - King's Mill Hospital, Sutton in Ashfield, Nottinghamshire
  - Barts Health NHS Trust - Whipps Cross University Hospital, London, Waltham Forest
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Baricitinib (LY3009104) in Participants With Rheumatoid Arthritis — https://trials.lillytrialguide.com/en-US/trial/4Pj7eUdQ6X850JMfBhUK23